CLINICAL TRIAL: NCT05051085
Title: "SpilleFri" - an Internet-delivered Treatment for Patients With Pathological Gambling. A Feasibility Pilot Study
Brief Title: Feasibility of the Internet-delivered Treatment "SpilleFri" for Patients With Pathological Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Westh Stenbro (Other)
Responsible Party: Sponsor-Investigator, Anna Westh Stenbro, Researcher, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-1-21
Record Dates: First submitted 2021-08-27; First posted 2021-09-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered treatment: "SpilleFri". (Experimental): All participants receive the internet-delivered therapist-assisted 8-modules treatment program "SpilleFri".
  Interventions: Behavioral: Internet-delivered treatment: "SpilleFri".

INTERVENTIONS:
Behavioral: Internet-delivered treatment: "SpilleFri". — The guided internet program consists of 8 modules over a period of 10 weeks. The content is written psychoeducation, videos with patients and experts, and exercises (encouraging reflection, cognitive restructuring, and exposure). The program is therapist-guided; hence all patients will receive support primarily from a specific therapist during the 10 weeks.

SUMMARY:
This uncontrolled feasibility pilot study explores the feasibility of a 10 week, 8-module, therapist-assisted, internet-delivered treatment program, "SpilleFri", for patients with Pathological Gambling. The study includes 25-30 participants aged 18-60 fulfilling diagnostic criteria for Pathological Gambling (ICD-10). The focus of the feasibility trial is evaluation of treatment response, treatment satisfaction, program utility, recruitment and retention rates, data completion rates, and time requirement. The primary feasibility criterion is 60 % of participants included in the study completing the treatment program.

DETAILED DESCRIPTION:
"SpilleFri" - an Internet-delivered Treatment for Patients with Pathological Gambling. A Feasibility Pilot Study

Lisbeth Frostholm & Anna Stenbro

Objective

The objective of this uncontrolled pilot study is to test the feasibility of a future RCT by exploring the feasibility of an internet-delivered treatment program, "SpilleFri", for patients with Pathological Gambling. The focus of the feasibility trial is evaluation of treatment response, treatment satisfaction, program utility, recruitment and retention rates, data completion rates, and time requirement. The primary feasibility criterion is an a priori defined change in patient-rated gambling problems from before to after treatment.

Design

This study is designed as an uncontrolled, single-arm, single-center feasibility pilot study.

Participants

The study includes 25-30 participants included from September 2021 to March 2022. The participants are recruited from The Research Clinic on Gambling Disorder, Aarhus University Hospital, Denmark. Patients with Pathological Gambling are screened for eligibility by the eligibility criteria below. They undergo thorough diagnostic assessment by an authorized psychologist including diagnostic interview (Schedules for Clinical Assessment in Neuropsychiatry).

Intervention

"SpilleFri" is a newly developed internet-delivered therapist-assisted treatment program for patients with Pathological Gambling. The 8 modules contain text, video files with psychoeducation, guided exercises, and videos with former patients. During a period of 10 weeks, patients are guided through the program modules assisted by a trained psychologist.

Course

If eligible and willing to participate, patients are included in the pilot study and assigned to a therapist (a trained psychologist from The Research Clinic on Gambling Disorder). Patients are contacted by telephone by the therapist and guided to login to the program platform and initiate treatment. The therapist follows the patient through the 8 treatment modules and provides guidance when needed. Patients and therapists primarily communicate through asynchronously written messages. If deemed necessary by the therapist, up to four consultations (telephone-/video-based or with physical attendance at the clinic) may be offered to enhance patient motivation and/or treatment adherence and effect. Treatment duration is 10 weeks.

Measurements

Patient-rated outcome measures are collected through a web-based program at the time of screening (before inclusion) (T1), before treatment (T2), and at end of treatment (T3). Between 6 and 12 patients will be interviewed during and post treatment to assess patient experience and satisfaction with the treatment program.

Clinician ratings are collected at the time of diagnostic assessment and at end of treatment.

Measurements also include logged data from the "SpilleFri"-treatment internet program, e.g. regarding patient activity in the program and number of messages to/from therapist pr. patient.

Feasibility outcomes

1. Recruitment and retention rates, time requirements and data completeness as measured by the rate of eligible patients willing to participate, the rate of included patients completing the treatment program (defined as completion of at least 5 modules), therapists' time spent per patient, and the rate of treatment completers providing full data
2. Patients' impression of treatment effect as measured by the clinical global improvement scale (CGI_p)
3. Patients' treatment satisfaction and assessment of program utility as measured by the credibility/expectancy questionnaire and a purpose designed patient satisfaction questionnaire
4. Therapists' impression of treatment effect as measured by the clinical global improvement scale (CGI_c).
5. Changes in patient-rated gambling problems from before to after the treatment measured by the NODS

Feasibility criteria

The investigators regard a future study testing the treatment program "SpilleFri" in an RCT as feasible if:

1. 60 % of the patients included in the study complete the treatment program (defined as completion of at least 5 of 8 modules)
2. 70 % of treatment completers provide data for primary gambling outcome variable (NODS)

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for Pathological Gambling (ICD-10)
* Able to read, wright, and speak Danish to a degree that enables interaction with the Danish internet treatment program, SpilleFri
* IT skills and access to internet and computer/tablet
* Willingness to participate in an internet-delivered psychological treatment program for Pathological Gambling

Exclusion Criteria:

* Current moderate or severe psychiatric disorder that demands special, individualized treatment, or clinical suspicion hereof, e.g. treatment-demanding depression, personality disorder, psychotic symptoms
* Untreated ADHD, ADD, or cognitive deficits that will most likely inhibit the patient from being able to read, understand, and work relatively independently in the SpilleFri internet program.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment and retention rate | Weekly during the intervention, up to 14 weeks
  Data will be gathered throughout the study to assess feasibility, defined herein as the extent to which the intervention can be successfully delivered.
  Primary feasibility outcome is recruitment and retention rate, collected through clinic records and therapist report in web-based questionnaire.

SECONDARY OUTCOMES:
Feasibility: Contact with therapist pr. patient | Weekly during the intervention, up to 14 weeks
  Collected through therapist report in web-based questionnaire and logged data from the treatment program "SpilleFri".
Feasibility: Patient activity in treatment program (log-in time and duration, yielding total minutes spend in treatment program) | Weekly during the intervention, up to 14 weeks
  Collected through logged data from the treatment program "SpilleFri"
Treatment expectancy and satisfaction | Immediately after inclusion in treatment. Before first treatment session
  Measured by the credibility/expectancy questionnaire. 6 items rated on a 1-9 or a 0%-100% scale, depending upon the item. The scale yields a mean expectancy score, ranging from maximum 100 % to minimum 0 %. Self-report collected through a web-based questionnaire program
Treatment expectancy and satisfaction | Immediately after the intervention
  Measured by the credibility/expectancy questionnaire. 6 items rated on a 1-9 or a 0%-100% scale, depending upon the item. The scale yields a mean satisfaction score, ranging from maximum 100 % to minimum 0 %. Self-report collected through a web-based questionnaire program
Clinician experience of treatment | Immediately after the intervention
  Qualitative and quantivative description of individual treatment courses including items measuring patient work effort, motivational barriers, amount of therapist quidance needed, and therapists' overall experience and satisfaction with working with the treatment program. Collected through questionnaire in web-based program.
Gambling problems past month, change | Baseline and immediately after the intervention
  Measured by Danish translation of The National Opinion Research Center Screen for Gambling Problems (NODS). 17 items with a maximum score of 10 (indicating a high level of gambling problems) and a minimum score of 0. Self-report measure collected through a web-based questionnaire program. For the purpose of the study, the NODS is modified to assess the last month instead of the last year.
  New versions of two NODS items are added, due to extensive clinical experience with two original NODS items being consistently misunderstood by patients (item 3 and 8).
Gambling behavior past week, change | Baseline (pre inclusion in treatment), post inclusion (before first session) and immediately after the intervention
  Purpose-made questionnaire with 6 items assessing present sense of control over gambling, gambling craving, motivation to stop gambling, and gambling behavior past week (including frequency, time spent, money spent, money won/lost). Self-report measure collected through a web-based questionnaire program. Each item is interpreted individually, yielding an indication of e.g. motivation to stop gambling ranging from 0 (low) to 2 (very high). Gambling frequency, money spent, and time spent is measured in respectively times pr. week, hours pr. week, Danish kroner pr. week)
Psychological well-being, change | Baseline and immediately after the intervention
  Measured on the Five Well-Being Index (WHO-5), a 5 item scale with a maximum score of 100 (indicating best imaginable well-being) and a minimum score of 0. Self-report collected through a web-based questionnaire program.
Stress, change | Baseline and immediately after the intervention
  Measured on two items from a stress assessment questionnaire developed by the Danish Health Authority ("Stress blandt unge", 2017). Self-report collected through a web-based questionnaire program.
Symptoms of anxiety, depression, and psychological distress, change | Baseline and immediately after the intervention
  Measured by 13 relevant subscores of the 92-item Danish version of the Symptom Checklist (SCL-92). All items are rated on 5point scales. Maximum and minimum scores for the items are respectively 20 and 4 for anxiety, 30 and 6 for depression, and 40 and 8 for general distress. Self-report collected through a web-based questionnaire program.
Overall health improvement | Immediately after the intervention
  Measured by the 5-point clinical global improvement scale (CGI). The CGI is measured by self-report (CGI_p) and by clinician rating (CGI_c). 1 item assessing overall improvement or worsening on a 5-point scale with a maximum score of 5 and a minimum score of 1. Self-report measure collected throguh a web-based questionnaire program.
Patient quality of life, change | Baseline and immediately after the intervention
  Measured on a 1 item, 11 point scale, where 10 indicates "the best possible life" and 0 indicates "the worst possible life". The scale is adapted from the Danish questionnaire "Ungdomsprofilen" from University of Southern Denmark. Self-report collected through a web-based questionnaire program.

CONTACTS AND LOCATIONS:
Overall Officials: Anna W Stenbro, MSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Research Clinic on Gambling Disorder (Forskningsklinikken for Ludomani), Funktionelle Lidelser, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Derived] Stenbro AW, Moldt S, Eriksen JW, Frostholm L. "I was Treated by the Program, the Therapist, and Myself": Feasibility of an Internet-Based Treatment Program for Gambling Disorder. J Gambl Stud. 2023 Dec;39(4):1885-1907. doi: 10.1007/s10899-023-10199-x. Epub 2023 Mar 31. PMID 37000310